CLINICAL TRIAL: NCT07078461
Title: Investigating the Safety and Efficacy of the 1927-nm Thulium Laser for Soft Tissue Coagulation in Keratosis Pilaris
Brief Title: Investigating the Safety and Efficacy of the 1927-nm Thulium Laser in Keratosis Pilaris
Acronym: KP
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Johns Hopkins University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: IRB00461291
Record Dates: First submitted 2025-07-21; First posted 2025-07-22 (Actual); Last update posted 2025-11-26 (Actual); Status verified 2025-11

CONDITIONS: Keratosis Pilaris (KP)
Keywords: keratosis pilaris; thulium; laser
MeSH Terms: conditions — Burnett Schwartz Berberian syndrome

STUDY DESIGN:
Intervention Model Description: Prospective cohort, open-label, split-body, randomized, single-blinded study
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (2):
- 1927-nm Thulium Laser therapy (right arm) (Active Comparator): Participants will receive treatment for Keratosis Pilaris with the 1927-nm Thulium laser on the right arm.
  Interventions: Device: 1927-nm Thulium Laser therapy
- 1927-nm Thulium Laser therapy (left arm) (Active Comparator): Participants will receive treatment for Keratosis Pilaris with the 1927-nm Thulium laser on the left arm.
  Interventions: Device: 1927-nm Thulium Laser therapy

INTERVENTIONS:
Device: 1927-nm Thulium Laser therapy — The investigators will use the LaseMD LEO Laser System (1927-nm Thulium laser) to create controlled, localized microscopic treatment zones (MTZs) of thermal injury to treatment area (unilateral upper arm). The investigators will utilize the random mode using the C1 tip (spot size 200 micrometers), which involves irradiation of the entire upper arm until diffuse erythema and edema appear. Additionally, the investigators may use the C5 tip (350 micrometers spot size) for focused treatment, up to five passes, until coagulation becomes evident. The maximum fluence for all C1 tip is 3-60 J/cm2 and 1-20 J/cm2 for C5 tips. The maximum pulse energy is 20 J with a pulse duration of 20 ms.

SUMMARY:
Keratosis pilaris (KP) is a very common skin condition that affects up to 80% of adolescents and 40% of adults. Clinically, KP causes rough dry patches and tiny spiny bumps around the hair follicles, as well as redness and pigmentation changes, most often on the upper arms, thighs, cheeks, or buttocks. While KP is benign, it can be cosmetically very bothersome. Currently, treatment options for KP are limited, and consist of topical moisturizers and keratolytic agents, but often leads to suboptimal improvements. In literature, many laser treatment modalities for KP have been studied, with varying results. The primary aim of this pilot study is to investigate how KP, a predominantly follicular disorder, responds to treatment with the 1927-nm Thulium laser.

DETAILED DESCRIPTION:
The non-ablative fractional 1927nm Thulium laser (LaseMD ULTRA) is approved by the Food and Drug Administration (FDA) for use in dermatological procedures requiring soft-tissue coagulation, such as treatment of actinic keratosis (pre-cancerous spots), and treatment of benign pigmented lesions such as, but not limited to lentigos (age spots), solar lentigos (sunspots) and ephelides (freckles). It is not approved for use for soft-tissue coagulation in keratosis pilaris.

It has been used in previous studies to treat conditions including acne scarring, skin rejuvenation, enlarged sebaceous glands, dyschromia, rosacea, and actinic keratoses. Its role as a potential treatment option for KP, remains unexplored.

ELIGIBILITY:
Inclusion Criteria:

* Female or male, in good health, ages 18-65
* Voluntarily signed informed consent form
* Any Fitzpatrick skin type (I-VI)
* Clinically diagnosed keratosis pilaris of bilateral upper arms
* Willing to have photographs taken and agree to the use of photographs for regulatory, presentation, or marketing purposes
* Willing and able to follow protocol procedures and requirements

Exclusion Criteria:

* History of receiving any laser therapy to the bilateral arms in the 12 months before recruitment
* History of or concurrent use of radiation to the bilateral arms in the 12 months before recruitment
* Participation of other device or drug clinical trials within 1 month before recruitment
* Concurrent diagnosis of active skin condition in the arms
* Presence of an active systemic or local skin disease that may affect wound healing
* History of forming keloids, collagen vascular disease, chronic drug or alcohol use
* History of malignant tumors in the upper arms
* Presence of open ulcers or infections any skin site
* Presence of a tan or sunburn over the upper arms in the month before recruitment
* Use of topical or oral photosensitizing medications
* Excessive body hair or tattoo in target area
* Pregnant and/or breastfeeding
* Presence of any medical conditions that interfere with subject's participation
* History of diagnosed pigmentary disorders in the target area
* Current smoker or history of smoking within 5 years

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 25 (Estimated)
Dates: Start 2025-10-23 (Actual); Primary Completion 2026-12 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Disease Severity as assessed by the Investigator's Global Assessment (IGA) | 6 weeks, 12 weeks, 18 weeks, 24 weeks, 2 follow up visits up to 3 months
  IGA score will be assessed by two blinded dermatologists for each arm based for two categories (erythema and texture/skin roughness) from standardized digital photographs. Scale ranges from 0 (clear) - 3 (severe). Lower score better.

SECONDARY OUTCOMES:
Global Improvement Scale (GIS) | 24 weeks, 2 follow up visits up to 3 months
  Global Improvement Scale (GIS) as rated by patients at last study visit and at follow-up visit(s). Scale range 0 (no improvement) - 4 (excellent improvement). Higher score better.
Participant Satisfaction | 24 weeks, 2 follow up visits up to 3 months
  Participant satisfaction rated from 0 (unsatisfied) - 3 (satisfied). Higher score more satisfaction.

CONTACTS AND LOCATIONS:
Overall Officials: Sarah Hsu, MD, Principal Investigator — Johns Hopkins University; Myriam Gonzalez, MD, Principal Investigator — Johns Hopkins University
Locations (1):
- Johns Hopkins University, Baltimore, Maryland, United States

REFERENCES:
- [Background] Weiss ET, Brauer JA, Anolik R, Reddy KK, Karen JK, Hale EK, Brightman LA, Bernstein L, Geronemus RG. 1927-nm fractional resurfacing of facial actinic keratoses: a promising new therapeutic option. J Am Acad Dermatol. 2013 Jan;68(1):98-102. doi: 10.1016/j.jaad.2012.05.033. Epub 2012 Oct 2. PMID 23041112
- [Background] Hassan AS, Abdel Aziz M, Saadi DG. Clinical and Dermoscopic Evaluation of Trichloroacetic Acid 20% Versus Long-Pulsed 1064-nm Nd-YAG Laser in the Treatment of Keratosis Pilaris. Dermatol Surg. 2022 Aug 1;48(8):838-842. doi: 10.1097/DSS.0000000000003488. Epub 2022 Jun 15. PMID 35917264
- [Background] Wong PC, Wang MA, Ng TJ, Akbarialiabad H, Murrell DF. Keratosis pilaris treatment paradigms: assessing effectiveness across modalities. Clin Exp Dermatol. 2024 Sep 18;49(10):1105-1117. doi: 10.1093/ced/llae066. PMID 38447098
- [Background] Wang MA, Wilson A, Murrell DF. A Review of the Scoring and Assessment of Keratosis Pilaris. Skin Appendage Disord. 2023 Aug;9(4):241-251. doi: 10.1159/000529487. Epub 2023 Apr 20. PMID 37564689